CLINICAL TRIAL: NCT05678673
Title: A Randomized Open-Label Phase 3 Study of XL092 + Nivolumab vs Sunitinib in Subjects With Advanced or Metastatic Non-Clear Cell Renal Cell Carcinoma
Brief Title: Study of XL092 + Nivolumab vs Sunitinib in Subjects With Advanced or Metastatic Non-Clear Cell Renal Cell Carcinoma
Acronym: STELLAR-304
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XL092-304; EU CTR: 2022-501703-27-0 (Other: European Medicines Agency)
Record Dates: First submitted 2022-12-23; First posted 2023-01-10 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Non-Clear Cell Renal Cell Carcinoma
MeSH Terms: interventions — Nivolumab; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- XL092 + Nivolumab (Experimental): Subjects with advanced or metastatic nccRCC will receive XL092 + nivolumab
  Interventions: Drug: XL092; Drug: Nivolumab
- Sunitinib Malate (Active Comparator): Subjects with advanced or metastatic nccRCC will receive an active comparator of sunitinib
  Interventions: Drug: Sunitinib Malate

INTERVENTIONS:
Drug: XL092 — Specified doses on specified days
  Arms: XL092 + Nivolumab
Drug: Nivolumab — Specified doses on specified days
  Other Names: Opdivo®
  Arms: XL092 + Nivolumab
Drug: Sunitinib Malate — Specified doses on specified days
  Other Names: Sutent®
  Arms: Sunitinib Malate

SUMMARY:
This is a multicenter, randomized (2:1), open-label, controlled Phase 3 trial of XL092 in combination with nivolumab versus sunitinib in subjects with unresectable, locally advanced or metastatic nccRCC who have not received prior systemic anticancer therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed nccRCC that is unresectable, advanced or metastatic. Histologic subtypes including papillary, unclassified, and translocation-associated are allowed. Among the eligible histologic subtypes, sarcomatoid features are allowed.
* Measurable disease according to RECIST v1.1 as determined by the Investigator.
* Available archival tumor biopsy material.
* Recovery to baseline or ≤ Grade 1 per CTCAE v5 from AE(s) related to any prior treatments unless AE(s) are deemed clinically nonsignificant by the Investigator and/or stable on supportive therapy.
* Age 18 years or older on the day of consent.
* Karnofsky Performance Status (KPS) ≥ 70%.
* Adequate organ and marrow function within 14 days prior to randomization.
* Sexually active fertile subjects and their partners must agree to use highly effective methods of contraception.
* Female subjects of childbearing potential must not be pregnant at screening.

Exclusion Criteria:

* Chromophobe, renal medullary carcinoma, and pure collecting duct histologic subtypes of nccRCC.
* Prior systemic anticancer therapy for unresectable locally advanced or metastatic nccRCC including investigational agents.

  * Note: One prior systemic adjuvant therapy, including immune checkpoint inhibitor therapy and excluding sunitinib, is allowed for completely resected RCC and if recurrence occurred at least 6 months after the last dose of adjuvant therapy.
* Radiation therapy for bone metastases within 2 weeks, any other radiation therapy within 4 weeks prior to randomization.
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy (including radiosurgery) or surgically removed and stable for at least 4 weeks before randomization.
* Concomitant anticoagulation with oral anticoagulants and platelet inhibitors. Subjects who are receiving oral anticoagulants at the time of screening must be transitioned to LMWH prior to randomization. Subjects who require treatment with platelet inhibitors are not eligible.
* Major surgery (eg, GI surgery, removal or biopsy of brain metastasis) within 8 weeks prior to randomization. Prior laparoscopic nephrectomy within 4 weeks prior to randomization. Minor surgery (eg, simple excision, tooth extraction) within 10 days before randomization. Complete wound healing from major or minor surgery must have occurred at least prior to randomization.

  * Note: Fresh tumor biopsies should be performed at least 7 days before randomization. Subjects with clinically relevant ongoing complications from prior surgical procedures, including biopsies, are not eligible.
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 480 ms per electrocardiogram (ECG) within 14 days before randomization.
* Pregnant or lactating females.
* Administration of a live, attenuated vaccine within 30 days before randomization.

  * Note: If feasible, approved non-live vaccines for SARS-CoV-2 should be administered at least 2 weeks before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Duration of Progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1), by Blinded Independent Radiology Committee (BIRC) | Approximately 27 months after the first subject is randomized
  Defined as the time from randomization to the earlier of either radiographic PD per RECIST 1.1 as determined by the BIRC or death from any cause
Objective response rate (ORR) as assessed by BIRC per RECIST 1.1 | Up to 24 months after the first subject is randomized
  Defined as the proportion of subjects with the best overall response of complete response (CR) or partial response (PR) per RECIST 1.1 as determined by the BIRC that is confirmed at a follow-up assessment ≥ 28 days later

SECONDARY OUTCOMES:
Duration of Overall Survival (OS) | Approximately 46 months after the first subject is randomized
  Defined as the time from randomization to death due to any cause

CONTACTS AND LOCATIONS:
Locations (163):
- United States (10):
  - Exelixis Clinical Site #1, Duarte, California
  - Exelixis Clinical Site #164, Newport Beach, California
  - Exelixis Clinical Site #162, San Francisco, California
  - Exelixis Clinical Site #163, Aurora, Colorado
  - Exelixis Clinical Site #55, Jacksonville, Florida
  - Exelixis Clinical Site #161, Buffalo, New York
  - Exelixis Clinical Site #58, New York, New York
  - Exelixis Clinical Site #15, New York, New York
  - Exelixis Clinical Site #42, Cleveland, Ohio
  - Exelixis Clinical Site #31, Dallas, Texas
- Argentina (6):
  - Exelixis Clinical Site #88, Pilar, Buenos Aires
  - Exelixis Clinical Site #89, Viedma, Río Negro Province
  - Exelixis Clinical Site #44, Buenos Aires
  - Exelixis Clinical Site #35, CABA
  - Exelixis Clinical Site #90, Córdoba
  - Exelixis Clinical Site #51, Santa Fe
- Australia (12):
  - Exelixis Clinical Site #94, Albury, New South Wales
  - Exelixis Clinical Site #97, Camperdown, New South Wales
  - Exelixis Clinical Site #98, Liverpool, New South Wales
  - Exelixis Clinical Site #95, Macquarie, New South Wales
  - Exelixis Clinical Site #92, Sydney, New South Wales
  - Exelixis Clinical Site #93, Waratah, New South Wales
  - Exelixis Clinical Site #99, Douglas, Queensland
  - Exelixis Clinical Site #100, Elizabeth Vale, South Australia
  - Exelixis Clinical Site #91, Box Hill, Victoria
  - Exelixis Clinical Site #96, St Albans, Victoria
  - Exelixis Clinical Site #14, Chermside
  - Exelixis Clinical Site #29, South Brisbane
- Brazil (12):
  - Exelixis Clinical Site #102, Porto Alegre, Rio Grande do Sul
  - Exelixis Clinical Site #68, Barretos
  - Exelixis Clinical Site #39, Itajaí
  - Exelixis Clinical Site #69, Passo Fundo
  - Exelixis Clinical Site #70, Porto Alegre
  - Exelixis Clinical Site #78, Porto Alegre
  - Exelixis Clinical Site #87, Santo André
  - Exelixis Clinical Site #50, São José do Rio Preto
  - Exelixis Clinical Site #101, São Paulo
  - Exelixis Clinical Site #81, São Paulo
  - Exelixis Clinical Site #85, São Paulo
  - Exelixis Clinical Site #43, São Paulo
- Bulgaria (3):
  - Exelixis Clinical Site #104, Plovdiv
  - Exelixis Clinical Site #105, Sofia
  - Exelixis Clinical Site #103, Sofia
- Chile (5):
  - Exelixis Clinical Site #53, Providencia
  - Exelixis Clinical Site #106, Santiago
  - Exelixis Clinical Site #108, Santiago
  - Exelixis Clinical Site #109, Santiago
  - Exelixis Clinical Site #107, Santiago
- Croatia (2):
  - Exelixis Clinical Site #111, Rijeka
  - Exelixis Clinical Site #110, Zagreb
- Czechia (4):
  - Exelixis Clinical Site #61, Brno
  - Exelixis Clinical Site #112, Olomouc
  - Exelixis Clinical Site #27, Prague
  - Exelixis Clinical Site #86, Prague
- Exelixis Clinical Site #71, Helsinki, Finland
- France (15):
  - Exelixis Clinical Site #115, Angers, Maine Et Loire
  - Exelixis Clinical Site #74, Caen
  - Exelixis Clinical Site #66, Clermont-Ferrand
  - Exelixis Clinical Site #40, Créteil
  - Exelixis Clinical Site #38, Le Mans
  - Exelixis Clinical Site #114, Lille
  - Exelixis Clinical Site #113, Lyon
  - Exelixis Clinical Site #36, Marseille
  - Exelixis Clinical Site #12, Paris
  - Exelixis Clinical Site #67, Paris
  - Exelixis Clinical Site #76, Pierre-Bénite
  - Exelixis Clinical Site #59, Reims
  - Exelixis Clinical Site #28, Rennes
  - Exelixis Clinical Site #41, Strasbourg
  - Exelixis Clinical Site #65, Suresnes
- Germany (3):
  - Exelixis Clinical Site #116, Frankfurt am Main, Hesse
  - Exelixis Clinical Site #79, Eisleben Lutherstadt
  - Exelixis Clinical Site #117, Hamburg
- Greece (6):
  - Exelixis Clinical Site #118, Athens
  - Exelixis Clinical Site #119, Athens
  - Exelixis Clinical Site #123, Athens
  - Exelixis Clinical Site #121, Thessaloniki
  - Exelixis Clinical Site #120, Thessaloniki
  - Exelixis Clinical Site #122, Tripoli
- Hong Kong (2):
  - Exelixis Clinical Site #124, Hong Kong
  - Exelixis Clinical Site #125, Hong Kong
- Hungary (3):
  - Exelixis Clinical Site #128, Budapest
  - Exelixis Clinical Site #127, Budapest
  - Exelixis Clinical Site #126, Debrecen
- Italy (14):
  - Exelixis Clinical Site #130, Rozzano, Milano
  - Exelixis Clinical Site #131, Candiolo, Torino
  - Exelixis Clinical Site #7, Arezzo
  - Exelixis Clinical Site #132, Bari
  - Exelixis Clinical Site #26, Brescia
  - Exelixis Clinical Site #19, Meldola
  - Exelixis Clinical Site #129, Milan
  - Exelixis Clinical Site #30, Napoli
  - Exelixis Clinical Site #37, Pavia
  - Exelixis Clinical Site #63, Pisa
  - Exelixis Clinical Site #48, Reggio Emilia
  - Exelixis Clinical Site #60, Roma
  - Exelixis Clinical Site #72, San Giovanni Rotondo
  - Exelixis Clinical Site #17, Verona
- Malaysia (3):
  - Exelixis Clinical Site #54, Kuala Lumpur
  - Exelixis Clinical Site #24, Kuala Lumpur
  - Exelixis Clinical Site #46, Putrajaya
- Exelixis Clinical Site #64, Eindhoven, Netherlands
- Poland (7):
  - Exelixis Clinical Site #45, Bydgoszcz
  - Exelixis Clinical Site #49, Gdansk
  - Exelixis Clinical Site #33, Otwock
  - Exelixis Clinical Site #77, Poznan
  - Exelixis Clinical Site #133, Poznan
  - Exelixis Clinical Site #80, Poznan
  - Exelixis Clinical Site #23, Rzeszów
- Exelixis Clinical Site #134, Singapore, Singapore
- Slovakia (3):
  - Exelixis Clinical Site #137, Banská Bystrica
  - Exelixis Clinical Site #135, Bratislava
  - Exelixis Clinical Site #136, Košice
- South Korea (13):
  - Exelixis Clinical Site #11, Busan
  - Exelixis Clinical Site #32, Busan
  - Exelixis Clinical Site #22, Daegu
  - Exelixis Clinical Site #13, Daejeon
  - Exelixis Clinical Site #16, Goyang-si
  - Exelixis Clinical Site #25, Gyeonggi-do
  - Exelixis Clinical Site #21, Seongnam-si
  - Exelixis Clinical Site #5, Seongnam-si
  - Exelixis Clinical Site #10, Seoul
  - Exelixis Clinical Site #4, Seoul
  - Exelixis Clinical Site #47, Seoul
  - Exelixis Clinical Site #6, Seoul
  - Exelixis Clinical Site #20, Seoul
- Spain (19):
  - Exelixis Clinical Site #143, Palma de Mallorca, Balearic Islands
  - Exelixis Clinical Site #142, Majadahonda, Madrid
  - Exelixis Clinical Site #56, Barcelona
  - Exelixis Clinical Site #9, Barcelona
  - Exelixis Clinical Site #52, Barcelona
  - Exelixis Clinical Site #138, Barcelona
  - Exelixis Clinical Site #141, Córdoba
  - Exelixis Clinical Site #62, Girona
  - Exelixis Clinical Site #139, Madrid
  - Exelixis Clinical Site #140, Madrid
  - Exelixis Clinical Site #3, Madrid
  - Exelixis Clinical Site #34, Madrid
  - Exelixis Clinical Site #8, Madrid
  - Exelixis Clinical Site #145, Málaga
  - Exelixis Clinical Site #57, Oviedo
  - Exelixis Clinical Site #75, Santander
  - Exelixis Clinical Site #144, Seville
  - Exelixis Clinical Site #18, Seville
  - Exelixis Clinical Site #73, Valencia
- Thailand (5):
  - Exelixis Clinical Site #147, Bangkok Noi, Bangkok
  - Exelixis Clinical Site #146, Phu Wiang, Changwat Khon Kaen
  - Exelixis Clinical Site #84, Bangkok
  - Exelixis Clinical Site #83, Bangkok
  - Exelixis Clinical Site #82, Chiang Mai
- Turkey (Türkiye) (10):
  - Exelixis Clinical Site #157, Adana
  - Exelixis Clinical Site #153, Adana
  - Exelixis Clinical Site #156, Ankara
  - Exelixis Clinical Site #149, Ankara
  - Exelixis Clinical Site #150, Ankara
  - Exelixis Clinical Site #155, Ankara
  - Exelixis Clinical Site #152, Ankara
  - Exelixis Clinical Site #151, Istanbul
  - Exelixis Clinical Site #148, Istanbul
  - Exelixis Clinical Site #154, Izmir
- United Kingdom (3):
  - Exelixis Clinical Site #158, Sheffield, South Yorkshire
  - Exelixis Clinical Site #160, London
  - Exelixis Clinical Site #159, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pal SK, Powles T, Kanesvaran R, Molina-Cerrillo J, Feldman DR, Barata P, Liu M, Bhatt A, Wang Z, Nandoskar P, Suarez C. STELLAR-304: a phase III study of zanzalintinib (XL092) plus nivolumab in advanced non-clear cell renal cell carcinoma. Future Oncol. 2025 Mar;21(7):787-794. doi: 10.1080/14796694.2025.2458395. Epub 2025 Feb 26. PMID 40008409